CLINICAL TRIAL: NCT05863078
Title: The Menus of Change Health and Heart Benefits for University Students (The MOCHAHS Trial): a Cross-sectional Study
Brief Title: The Menus of Change Health and Heart Benefits for University Students
Status: Not yet recruiting | Type: Observational
Sponsor: University of Reading (Other)
Responsible Party: Principal Investigator, Charlotte E Mills, Principle Investigator, University of Reading
Other Study IDs: TBC
Record Dates: First submitted 2023-02-08; First posted 2023-05-17 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Healthy Lifestyle
Keywords: Menus of Change; Arterial stiffness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood and urine samples will be taken from participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group following the Menus of Change diet
- Group not following the menus of Change diet

SUMMARY:
The goal of this cross-sectional study is to investigate the health benefits of the Menus of Change in undergraduate university students, by comparing 2 groups: Students eating in the Menus of change catered halls, versus students eating outside the Menus of change meal plan. The main question it aims to answer is:

What are the effects of the menus of change on other vascular outcomes, namely blood pressure? What are the effects of the menus of change on other health markers?

DETAILED DESCRIPTION:
The Menus of Change (MoC) is an example of behaviour change that was created by The Culinary Institute of America (CIA) and Harvard TH Chan School of Public Health. This initiative is based on a set of around 24 core principles, mainly promoting and serving 'healthy, sustainable, and delicious' food in restaurants and foodservice operations. The University of Reading has successfully implemented the MoC across the campus and in students' accommodations. However, MoC is not implemented across all campus halls.

To date, most of the studies performed in relation to the MoC had explored techniques to encourage students towards healthier, more sustainable diets. Very little research focuses on the associated health outcomes and hence the impact on health of the eating pattern laid out in the MoC principles.

Therefore, this project aims to investigate the health impact of the menu of change on university students, by comparing 2 groups: students eating in MoC catered halls, following the meal plan provided by the university food services, versus students who do not follow the menus of change meal plan. The primary aim will be to investigate the effect of the MoC on vascular outcomes, namely arterial stiffness, a particularly important tool in younger adults with low-moderate cardiovascular disease risk.

Secondary aims will be to investigate other vascular outcomes, namely blood pressure changes, as well as looking at other health markers, such as full blood count, lipid profile, sugar levels, liver and kidney function, and CVD related inflammatory markers. In addition, the study aims to look at the impact of the MoC on stress and anxiety levels and the differences in students' attainment between groups.

ELIGIBILITY:
Inclusion Criteria:

* Adults
* Home students living in university halls
* Undergraduates
* Can understand participant information sheet and willing to comply with the study design

Exclusion Criteria:

* International students
* postgraduates
* living outside the university halls
* participating in other studies

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants eating in the university halls following the Menus of Change diet will be selected and compared to participants living in the university halls but not following the Menus of Change and therefore eating outside the university dining halls
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Arterial stiffness | up to 2 weeks after completing a 3-day food diary
  Arterial stiffness will be measured using Mobil-O-Graph to assess the cardiovascular risk in participants

SECONDARY OUTCOMES:
Full blood count | up to 2 weeks after completing a 3-day food diary
  Full blood count levels will be compared between both groups
Lipid profile | up to 2 weeks after completing a 3-day food diary
  Lipid profile levels will be compared between both groups
Glucose levels | up to 2 weeks after completing a 3-day food diary
  by comparing levels between both groups
liver profile | up to 2 weeks after completing a 3-day food diary
  comparing liver profile levels between both groups
Kidney profile | up to 2 weeks after completing a 3-day food diary
  kidney profile levels to be compared between both groups
SCFA levels | up to 2 weeks after completing a 3-day food diary
  short chain fatty acids levels to be compared between both groups
Cardiovascular disease related inflammatory biomarkers | up to 2 weeks after completing a 3-day food diary
  Levels to be compared between both groups

OTHER OUTCOMES:
Depression and anxiety survey | up to 2 weeks before the study visit
  Beck's depression survey, STAI 1 and PANAS
Academic attainment | By the end of academic year
  To assess the relationship between healthy diet and academic results
Urine dietary biomarkers level | 24-hours before the study visit
  by 24-hours urine sample

IPD SHARING:
Plan to Share IPD: Undecided